CLINICAL TRIAL: NCT07076394
Title: The Effects of Forgiveness Education
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-1790; A173000 (Other: UW Madison); Protocol Version 12/2/24 (Other: UW Madison)
Record Dates: First submitted 2025-07-14; First posted 2025-07-22 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Forgiveness

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Forgiveness Education (Experimental): classes delivered once a week for 12 weeks
  Interventions: Behavioral: Forgiveness Education
- Control Group (No Intervention)

INTERVENTIONS:
Behavioral: Forgiveness Education — The curriculum will apply the textbook of "Forgiveness is a Choice: A Step-by-Step Process for Resolving Anger and Restoring Hope" written by Dr. Robert Enright.
  Arms: Forgiveness Education

SUMMARY:
This study aims to investigate the effects of forgiveness education.

DETAILED DESCRIPTION:
Participation in this study will contribute to promoting the physical and mental health of college school students, improving their quality of life, and maintaining campus and online security.

The intervention program involved in this study is to better psychological welfare.

The number of questionnaires at each testing time is 9 (pre-intervention test only has 7 questionnaires to fill in due to previously completed 2 questionnaires in the eligibility survey), and the approximate length of time it will take to complete the scales is around 40 minutes

ELIGIBILITY:
Inclusion Criteria:

* first and second year college students at Changzhi Preschool Teachers College

Exclusion Criteria:

-

Ages: 19 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2025-09-08 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Flourishing Scale Score | pre-intervention (baseline), post-intervention (12 weeks on study), follow-up (16 weeks on study)
  8-items scored on a 7 point likert scale from 1 (strongly disagree) to 7 (strongly agree) for a total possible range of scores from 8 to 56 where higher scores demonstrate a person with many psychological resources and strengths.
Social Desirability Scale Score | pre-intervention (baseline), post-intervention (12 weeks on study), follow-up (16 weeks on study)
  33-item true or false survey where the score is the sum of statements assessed to be true. Scores range from 0-33, where higher scores indicate higher social desirability.
Rosenberg Self-Esteem Scale Score | pre-intervention (baseline), post-intervention (12 weeks on study), follow-up (16 weeks on study)
  10-item measure scored from 1 (strongly agree) to 4 (strongly disagree). After accounting for several reverse-scored items, scores are summed from 10 to 40, higher scores indicate higher self-esteem.
PROMIS Emotional Distress - Anger Score | pre-intervention (baseline), post-intervention (12 weeks on study), follow-up (16 weeks on study)
  5-item survey scored from 1 (never) to 5 (always) for a range of scores from 5 to 25 where higher scores indicate increased anger.
PROMIS Emotional Distress - Anxiety Score | pre-intervention (baseline), post-intervention (12 weeks on study), follow-up (16 weeks on study)
  8-item survey scored from 1 (never) to 5 (always) for a range of scores from 8 to 40 where higher scores indicate increased anxiety.
Herth Hope Index Score | pre-intervention (baseline), post-intervention (12 weeks on study), follow-up (16 weeks on study)
  12-item survey, scores range from 12 to 48 where higher scores indicate higher hope.
Enright Forgiveness Inventory (EFI-30) Short Form Score | pre-intervention (baseline), post-intervention (12 weeks on study), follow-up (16 weeks on study)
  EFI-30 surveys 3 subscales for forgiveness: affective, behavioral, cognitive. It is scored from 1 (strongly disagree) to 6 (strongly agree), total scores range from 30-180, where higher scores indicate increased levels of forgiveness.
*Peer Influences Scale Score | pre-intervention (baseline), post-intervention (12 weeks on study), follow-up (16 weeks on study)
  18-item survey scored from 0-4, total range of scores from 0-72. *Scale will be identified and further clarified after study is complete to preserve study integrity.
*Peer Influences Scale Score II | pre-intervention (baseline), post-intervention (12 weeks on study), follow-up (16 weeks on study)
  16-item survey scored from 0-6, total range of scores from 0-96. *Scale will be identified and further clarified after study is complete to preserve study integrity.

CONTACTS AND LOCATIONS:
Overall Officials: Robert D Enright, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- Changzhi Preschool Teachers College, Changzhi, Shanxi, China

IPD SHARING:
Plan to Share IPD: No